CLINICAL TRIAL: NCT03441659
Title: Anterior Cruciate Ligament Reconstruction: Clinical Outcome at Middle and Long Term Follow-Up
Brief Title: ACL Reconstruction: Clinical Outcome
Acronym: RIC-ACL
Status: Recruiting | Type: Observational
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Prof, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 0007043
Record Dates: First submitted 2017-08-29; First posted 2018-02-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-06

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ACL reconstruction — Surgical ACL reconstruction

SUMMARY:
The study is intended to include all patients who will undergo surgical reconstruction of the anterior cruciate ligament (ACL). The patients will be monitored and evaluated preoperatively and also at 6 months and 1, 2 and 5 years after the intervention through a clinical visit or telephone interview. Such assessments will include the administration of questionnaires to determine the patient's functional symptoms and the objective examination of the knee during a medical examination to quantify its stability.

DETAILED DESCRIPTION:
The literature presents a number of studies on the reconstruction of the anterior cruciate ligament, as well as numerous registers, but the identification of factors and parameters determining the clinical outcomes remains largely debated. The study aims to offer new elements to analyze this treatment and potentially identify the factors responsible for the outcomes and the factors useful to optimize the clinical outcome in the future. In fact, in addition to collect patient data in terms of features and clinical-functional status, objective data will be documented and correlated. In particular the quantification of knee laxity will be performed using an innovative device based on the use of inertial sensors (a methodology recently developed and already validated at the Istituto Ortopedico Rizzoli). The study is intended to include all patients who will undergo surgical reconstruction of the anterior cruciate ligament (ACL). These patients will be followed and evaluated preoperatively, at 6 months and at 1, 2 and 5 years after surgery during a clinical visit or a telephone interview. Such evaluations will include the submission of questionnaires to determine the patient's functional symptoms and also knee joint assessment during a medical examination to quantify the knee joint stability.

Moreover, the following clinical scores will be adopted: IKDC-subjective, IKDC-objective, SF12, Marxs, Koos, Tegner, VAS for pain assessment, EQ-VAS for overall health status assessment. Also it will be recorded the lapse of time for returning to work and sports, the degree of patient satisfaction,the adverse events, the failures and any new treatments on the same site.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have provided informed written written consent;
2. Patients aged between 18 and 60;
3. Patients undergoing reconstructive surgical treatment of the anterior cruciate ligament (ACL)

Exclusion Criteria:

1. Patients unable to understand and to want;
2. Patients who have not signed informed consent;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ACL lesions and undergoing to surgical ACL reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Knee Laxity Assessment | 5 years
  Laxity Evaluation with KiRA device

SECONDARY OUTCOMES:
SF12 Score | 5 years
  The SF-12v2 is an abbreviated version of the SF-36. SF-36 is the best-known and most widely used measure of health-related quality of life in the international literature. It measures different health concepts through 36 multiple-choice questions, data are aggregated into 8 scales investigating: physical activity, role and physical health, physical pain, Health in general, vitality, social activities, role and emotional state, mental health, a question on change in health status during the last year is also added.
Marx Activity Rating Score | 5 years
  The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year.
KOOS Score | 5 years
  KOOS SCORE consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items).
  Each question is scored from 0 to 4, where 0 indicates "no difficulty" and 4 "severe difficulty. Score range 0-100 for each subscale
IKDC Score | 5 years
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function.
VAS Score | 5 years
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable"

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Zaffagnini, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: No